CLINICAL TRIAL: NCT02886273
Title: DIagnostics, RBC Levels of n-3 Fatty Acids and Serum Vitamin D in Patients With Out-of-Hospital Cardiac Arrest (OHCA)
Brief Title: DIagnostics, Fatty Acids and Vitamin D in SCA
Acronym: DIFAD-SCA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Helse Stavanger HF (Other Government)
Responsible Party: Sponsor
Other Study IDs: StavangerSCA
Record Dates: First submitted 2016-08-23; First posted 2016-09-01 (Estimated); Last update posted 2021-08-11 (Actual); Status verified 2021-01

CONDITIONS: Out-of-Hospital Cardiac Arrest; Ventricular Fibrillation
Keywords: Sudden Cardiac Arrest; Out-of-hospital; Ventricular fibrillation; Classification; Mechanisms; Biomarkers
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Ventricular Fibrillation; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples Without DNA — 20 ml of EDTA-blood for preparation of red blood cells and plasma will be harvested during resuscitation or immediately after return of spontaneous circulation (ROSC) from a peripheral venous catheter (PVC) or arterial line. After hospital admission blood samples will be collected from survivors according to general routines at our hospital. For survivors an extra set of blood samples consisting of 6 ml EDTA-blood, 6 ml citrate-blood and 6 ml serum will be taken after 8-12 hours and 24-48 hours.
  All blood samples taken at inclusion will be immediately centrifuged and stored in aliquots at - 70o C until the measurements can be performed. Laboratory technicians will be blinded with respect to clinical data.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Group 1: SCA with first MI (n = 43)
  Interventions: Other: Group 1
- Group 2: SCA with AMI and previous MI (n = 10)
  Interventions: Other: Group 2
- Group 3: SCA without AMI and without former heart disease (n = 3)
  Interventions: Other: Group 3
- Group 4: SCA without AMI and with known heart disease (n = 18)
  Interventions: Other: Group 4

INTERVENTIONS:
Other: Group 1 — Observation
  Groups: Group 1
Other: Group 2 — Observation
  Groups: Group 2
Other: Group 3 — Observation
  Groups: Group 3
Other: Group 4 — Observation
  Groups: Group 4

SUMMARY:
Sudden cardiac death (SCD) is a major cause of mortality in industrialized countries and represents a major health issue. The survival rate after out-of-hospital cardiac arrest (OHCA) is only 10-15%, regardless of first recorded rhythm. Prior heart disease is a major risk factor for sudden cardiac arrest (SCA), and coronary artery disease (CAD) is the most common underlying cause. A better understanding of pathophysiological mechanisms occurring during cardiac arrest (CA), earlier diagnosis of underlying cause as well as identification of risk factors related to CA may improve patient treatment and increase survival. In our out-of-hospital cardiac arrest (OHCA)-study, we intend to investigate whether biomarkers, such as copeptin, hs-cTnT and NT-proBNP in addition to clinical evaluation may improve risk stratification and supply information related to pathophysiology.

Furthermore, we intend to gather additional pathophysiological information related to coagulation activation in CA and cardiopulmonary resuscitation (CPR), as intravascular thrombosis may impair microcirculation and reduce end-organ blood flow which is associated with a poor prognosis. We intend to study coagulation activation during and immediately after SCA with regard to outcome, and assess the contribution of the intrinsic system, measured together with that of the extrinsic system.

Low levels of n-3 fatty acids (FA) are reported as a risk factor for SCD. Red blood cell eicosapentaenoic acid (EPA) + docosahexaenoic acid (DHA) may serve as a useful surrogate of cardiac omega-3 fatty acid status. The exact mechanism by which FAs might protect against serious cardiac arrhythmias is not known, but they are expected to exert a membrane stabilizing effect during an ischemic episode. In our study we intend to evaluate the association between ventricular fibrillation (VF) and the content of EPA and DHA in red blood cells. Furthermore, as vitamin D is associated with n-3 FAs in the diet, we also aim at investigating the association between 25-hydroxy (OH)-vitamin D and VF.

DETAILED DESCRIPTION:
Background:

Sudden cardiac death (SCD), also termed sudden cardiac arrest (SCA), accounts for approximately 15 percent of the total mortality in industrialized countries. In Europe, the incidence of out-of-hospital Emergency Medical Services (EMS) attended sudden cardiac arrest (SCA) is estimated to 81.6/100 000 person-years, 52.5 % of which is presumed to have a cardiac cause [1]. Coronary artery disease (CAD) is the most common underlying heart disease associated with out-of-hospital cardiac arrest (OHCA) [2]. SCD is the initial presentation of CAD in 15 percent of CAD-patients [3]. Furthermore, it is also the most frequent mechanism of death in patients with known CAD, accounting for 40-50 percent of CAD-mortality [4]. Compared to healthy subjects the incidence of SCD is six- to tenfold higher in the presence of clinically recognized heart disease [5], and cardiomyopathies represents the second largest cause of SCD [6]. Despite early advanced cardiopulmonary resuscitation (CPR) provided by the EMS the mortality rate remains high [1]. Due to the dramatic consequence of SCA, understanding of pathophysiological mechanisms and early identification of etiology is essential to improve outcome.

SCA due to VF may be the presenting symptom of acute myocardial ischemia or may be a consequence of scarring due to a previous myocardial infarction (MI). Cardiac troponin (c-Tn) is the most commonly used biomarker for diagnosing an acute myocardial infarction (AMI) [7]. Although earlier detection of AMI may be obtained by the introduction of high sensitivity (hs)-cTn assays, there still remains a troponin-blind period very early after symptom onset [8, 9], with the need for serial blood sampling to diagnose or exclude an AMI [7, 9]. Furthermore, there are challenges related to the specificity of elevated levels of hs-cTn [10, 11]. Therefore, measurement of hs-cTn in a single blood draw in the ambulance or at admission may not provide sufficient information for the diagnosis of AMI among patients with OHCA.

Lately, several studies have demonstrated an incremental diagnostic value of copeptin when added to conventional cTn or hs-cTn for early detection of AMI [12, 13]. Copeptin levels peak early (0-1 h) after symptom onset and are already increased at the time of first medical contact in the ambulance for patients with MI [8]. Copeptin used in combination with hs-cTn may therefore improve the diagnosis of AMI in very early presenters, and help differentiating the underlying cause of SCD.

Copeptin has also been demonstrated to be an independent predictor of adverse events following MI [14] and is shown to be associated with outcome after OHCA [15, 16]. Less is known about the prognostic value of troponins in patients experiencing a cardiac arrest (CA). Higher values of hs-cTnT are seen in one-year non-survivors as compared to survivors of OHCA, although not shown to be an independent predictor of 12-months survival [10]. In our study, the objective will be to evaluate the diagnostic and prognostic utility of hs-cTnT and copeptin in SCA patients.

Patients with heart failure are at increased risk for ventricular arrhythmias and SCD. B-type natriuretic peptide (BNP) and N-terminal proBNP (NT-proBNP) have been demonstrated to be useful diagnostic tools to rule out both chronic and acute heart failure [17]. Little is known about the natural course of natriuretic peptides during a SCA event, but BNP is demonstrated to be an independent predictor of long-term mortality [18], as well as survival to hospital discharge after OHCA of cardiac origin [19]. There is also a well-documented association between BNP or NT-proBNP and the short- and long-term risk of death in patients with acute coronary syndrome (ACS) [20, 21]. In our study, we intend to investigate the diagnostic and prognostic utility of NT-proBNP sampled during or immediately after OHCA.

The overall survival rate after OHCA is low. Even in successfully resuscitated patients admitted to the intensive care unit (ICU), the prognosis remains poor. Former studies have shown a marked activation of blood coagulation, with a concomitant inadequate activation of the endogenous fibrinolytic system, in resuscitated OHCA-patients [22-25]. Intravascular clotting and "no reflow" in the microvasculature represent a barrier to successful end-organ perfusion and may influence the outcome in cardiac arrest (CA) patients [26]. Understanding the pathophysiological mechanisms of CA is important to guide management and improve outcome. Plasma thrombin-antithrombin (TAT) complexes, fibrin monomers (FM) and D-dimer are used as specific markers of activated blood coagulation. Previous studies have shown markedly increased TAT-levels in patients with nontraumatic OHCA [22, 23]. Admission TAT is also shown to be a useful prognostic marker in resuscitated OHCA patients and is independently associated with survival after resuscitation from CA [24]. D-dimer levels are found to increase after CA and CPR [22, 27]. Accordingly, Adrie et al. [28] demonstrated high admission levels of D-dimer in all OHCA patients. Furthermore Szymanski et al. [29] reported higher D-dimer concentrations on admission to be a strong and independent predictor of mortality in OHCA patients. In our study, we intend to study the activation of blood coagulation, including both the extrinsic- and the intrinsic coagulation pathways, during and immediately after SCA with regard to outcome.

Most interventions to date do not directly affect the transient pathophysiologic event initializing potentially fatal arrhythmias. Instead, they attempt to alter and prevent underlying disease like CAD. Animal studies have shown that fish oils are protective against ischemia-induced VF [30]. Support for these data comes from the Physicians' Health Study [31], which is a prospective study of 20 551 men aged 40 to 84, free of cardiovascular disease at baseline, with a follow-up period of 11 years. As compared to consumption of fish less than once a month, fish intake at least once per week was associated with a reduced risk of SCD (RR 0.48). In the same study there was no reduction in the risk of total myocardial infarction, non-sudden cardiac death or total cardiovascular mortality, and the protective effect of fish was suggested to be due to a reduction in fatal ventricular arrhythmias. It has been hypothesized that the lower risk of SCD with higher fish intake may be related to the long-chain n-3 polyunsaturated fatty acids (PUFAs) EPA and DHA found in fish. Consistent with this hypothesis are the observations from the physicians' Health Study [31] that the risk of SCD was significantly lower in subjects with blood n-3 FA levels in the highest as compared to the lowest quartile. The same potential effect of fish oils to protect against SCD was illustrated in the randomized, open-controlled GISSI-prevention study [32]. Patients with a recent myocardial infarction receiving n-3 FAs supplements had a significant lower incidence in the combined endpoint of death plus nonfatal infarction and nonfatal stroke at 42 months (12.6 versus 13.9%). After adjustment for risk factors, all of the observed benefit was due to a 20 % reduction in the risk of death, mostly due to reduction in SCD. However, a study of 200 patients secured with an ICD (implantable cardioverter defibrillator) following an episode of ventricular tachycardia (VT) or VF, has not shown a reduction in the recurrence of these arrhythmias after supplementation with EPA/DHA. In that study there was actually a trend toward a higher incidence of VT/VF in patients randomized to EPA/ DHA substitution [33]. In that setting the underlying mechanism for the generation of VF might, however, not be ischemic.

The exact mechanism by which FAs might protect against serious cardiac arrhythmias is not known. They are important constituents of cell membranes and may affect several electrophysiologic properties, such as resting potential, action potential, repolarization and refractory period. Alterations in cellular calcium concentration can contribute significantly to changes in both impulse generation and impulse conduction in myocardial cells. Incorporation of n-3 fatty acids in the cellular membrane is shown to affect membrane fluidity which in turn may have an influence on calcium entry or removal. An alternative mechanism may be changes effected by n-3 FAs on myocardial production of eicosanoids. In particular the inhibition of thromboxane A2 (TXA2) production is likely to be of significant pathophysiological benefit, since TXA2 is shown to be implicated in myocardial ischemia and arrhythmogenesis [34].

A recent study by William S. Harris et al. [35] has shown that levels of EPA/ DHA in cell membranes of red blood cells (RBC EPA/ DHA) highly correlate with the cardiac EPA/ DHA level. The RBC response to supplementation was also very similar to that observed in the heart. Therefore RBC EPA+ DHA may serve as a useful surrogate of cardiac omega-3 fatty acid status. The investigators expect n-3 FAs to exert a membrane stabilizing effect during an ischemic episode, and hypothesize that patients suffering VF during the initial phase of their first AMI presentation have lower levels of RBC EPA/ DHA than matched controls.

Over the last years vitamin D is another dietary supplement found to be associated with cardiovascular disease. This fat-soluble vitamin, primarily derived from sun-exposure and fatty fish, has been demonstrated to influence cardiac contractility and myocardial calcium homeostasis [36], and insufficiency of this vitamin may have deleterious effects on cardiac autonomic functions as evaluated by heart rate turbulence and heart rate variability [37]. In prospective studies, severe vitamin D deficiency has been strongly associated with total mortality, cardiovascular events and SCD [38-42]. In one study of 3299 patients who were routinely referred to coronary angiography, the authors demonstrated hazard ratios for death due to heart failure and for SCD of 2.84 (1.20-6.74) and 5.05 (2.13-11.97), respectively, when comparing patients with severe vitamin D deficiency [25(OH)D <25 nmol/liter)] with persons in the optimal range [25(OH)D ≥ 75 nmol/liter] [43]. Demonstrated effects on electrophysiology,contractility, and cardiac structure suggest that vitamin D deficiency might actually be a causal factor for development of cardiac diseases. The pronounced effect on SCD found in several studies might be an indication of a possible protective effect of high vitamin D-levels against ventricular arrhythmias. This is, however, not well studied and the optimal cut-off-value for protection is not well defined. Therefore, a comparison of the 25-OH-vitamin D levels between different OHCA categories of patients, with and without an acute coronary event, may be appropriate.

Statistical methods

Statistical analysis will be performed using the statistical package SPSS (Statistical Package for the Social Sciences). A statistically significant level of p < 0.05 will be applied for all tests.

EPA/ DHA and vitamin D in the different clinical patient categories will be compared to controls collected from the RACS (Risk markers in the Acute Coronary Syndromes) database (NCT00521976).

Ethics and confidentiality

The present study is conducted in accordance with the Helsinki Declaration of 1975 and later revisions and accepted by the Regional Board of Research Ethics as well as the Norwegian Health Authorities. Analytic data will be related to patient number and not to patient identity. According to Norwegian regulations, the family of non-survivors will be informed by the attending physician and the inclusion of patients needs to be documented in the hospital records. The family of the deceased is entitled to object to the use of any biological samples for research purposes. Patients regaining consciousness and mental capability during their hospital stay will be asked personally for a written informed consent. For the remaining survivors the next of kin will be asked for permission on behalf of the patient. If either the patient or the family refuses participation, blood samples already collected at resuscitation and admission will be destroyed.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. OHCA of assumed cardiac etiology
3. Documented first recorded heart rythm

Exclusion Criteria:

1. Evidence of non-cardiac death (including cerebral etiology and pulmonary embolism)
2. OHCA due to cardiac tamponade.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recruitment:
  Patients with Out-of Hospital Cardiac Arrest (OHCA) of assumed cardiac origin will be recruited by the ambulance emergency team.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2007-01 (Actual); Primary Completion 2010-12 (Actual); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Early diagnostic performance of copeptin in Out-of-Hospital Cardiac arrest (OHCA) due to ventricular fibrillation (VF) | 48 hours
  Comparison with high sensitivity cardiac Troponin T.

SECONDARY OUTCOMES:
EPA and DHA as compared to other fatty acids in red blood cell membranes from patients with OHCA | 48 hours
  Applying matched controls
25-hydroxy (OH)-vitamin D in subjects with OHCA due to ventricular fibrillation (VF) | 48 hours
  Applying matched controls
Survival rate in OHCA with documented ventricular fibrillation | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Dennis WT Nilsen, MDd PhD, Principal Investigator — Helse Stavanger HF
Locations (1):
- Stavanger University Hospital, Stavanger, Rogaland, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aarsetoy R, Omland T, Rosjo H, Strand H, Lindner T, Aarsetoy H, Staines H, Nilsen DWT. N-terminal pro-B-type natriuretic peptide as a prognostic indicator for 30-day mortality following out-of-hospital cardiac arrest: a prospective observational study. BMC Cardiovasc Disord. 2020 Aug 24;20(1):382. doi: 10.1186/s12872-020-01630-x. PMID 32838754
- [Result] Aarsetoey H, Aarsetoey R, Lindner T, Staines H, Harris WS, Nilsen DW. Low levels of the omega-3 index are associated with sudden cardiac arrest and remain stable in survivors in the subacute phase. Lipids. 2011 Feb;46(2):151-61. doi: 10.1007/s11745-010-3511-3. Epub 2011 Jan 14. PMID 21234696
- [Result] Aarsetoy R, Aarsetoy H, Hagve TA, Strand H, Staines H, Nilsen DWT. Initial Phase NT-proBNP, but Not Copeptin and High-Sensitivity Cardiac Troponin-T Yielded Diagnostic and Prognostic Information in Addition to Clinical Assessment of Out-of-Hospital Cardiac Arrest Patients With Documented Ventricular Fibrillation. Front Cardiovasc Med. 2018 Jun 7;5:44. doi: 10.3389/fcvm.2018.00044. eCollection 2018. PMID 29930943
- [Derived] Aarsetoy R, Ten Cate H, Spronk H, Van Oerle R, Aarsetoy H, Staines H, Nilsen DWT. Activated factor XI-antithrombin complex presenting as an independent predictor of 30-days mortality in out-of-hospital cardiac arrest patients. Thromb Res. 2021 Aug;204:1-8. doi: 10.1016/j.thromres.2021.05.014. Epub 2021 May 29. PMID 34089982